CLINICAL TRIAL: NCT03571750
Title: "Building Stronger Allies": Development and Evaluation of a Web Application Targeting Interpersonal Risk Factors for Suicide in Active Duty Service Members
Brief Title: Building Stronger Allies
Acronym: BSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: W81XWH-16-2-003
Record Dates: First submitted 2018-05-21; First posted 2018-06-28 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Suicide; Risk Reduction
Keywords: Suicide; Prevention; Risk Factor; Intervention; Military
MeSH Terms: conditions — Suicide; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Approximately 510 participants will be randomly assigned to one of two conditions (1) BSA or (2) HET Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Building Stronger Allies Condition (Experimental): BSA was developed to model the educational and behavioral techniques commonly employed in the treatment of individuals with mood psychopathology. The psychoeducation portion uses Cognitive Behavioral Therapy principles to correct problematic ideas and behaviors related to PB/TB. More specifically, the program was designed to correct "myths" regarding PB/TB. The program emphasizes the idea that social interaction is a critical need, just like other basic needs such as the need for food and water. Participants are taught that negative beliefs about being isolated and being a burden are usually inaccurate. Following this, behavioral activation techniques are introduced as a way to decrease isolation and feelings of burdensomeness.
  Interventions: Behavioral: Building Stronger Allies
- Health Education Training Condition (Placebo Comparator): In the HET condition, participants will spend approximately the same amount of time with a program that will present information regarding the importance and benefits of a maintaining a healthy lifestyle and then will provide guidelines to achieve a healthy lifestyle. HET is shown to engage participants with beneficial information while being inert with respect to the risk mechanisms of interest (i.e., PB/TB). The program covers a number of health related topics including: diet, alcohol use, water consumption, exercise, and sleep. The program reviews with the Participants how to monitor their own daily health habits, which will be reinforced by the Smartphone application.
  Interventions: Behavioral: Health Education Training

INTERVENTIONS:
Behavioral: Building Stronger Allies — BSA was developed to model the educational and behavioral techniques commonly employed in the treatment of individuals with mood psychopathology. The psychoeducation portion uses Cognitive Behavioral Therapy principles to correct problematic ideas and behaviors related to PB/TB. More specifically, the program was designed to correct "myths" regarding PB/TB. The program emphasizes the idea that social interaction is a critical need, just like other basic needs such as the need for food and water. Participants are taught that negative beliefs about being isolated and being a burden are usually inaccurate. Following this, behavioral activation techniques are introduced as a way to decrease isolation and feelings of burdensomeness.
  Other Names: BSA
  Arms: Building Stronger Allies Condition
Behavioral: Health Education Training — In the HET condition, participants will spend approximately the same amount of time with a program that will present information regarding the importance and benefits of a maintaining a healthy lifestyle and then will provide guidelines to achieve a healthy lifestyle. HET is shown to engage participants with beneficial information while being inert with respect to the risk mechanisms of interest (i.e., PB/TB). The program covers a number of health related topics including: diet, alcohol use, water consumption, exercise, and sleep. The program reviews with the Participants how to monitor their own daily health habits, which will be reinforced by the Smartphone application.
  Other Names: HET
  Arms: Health Education Training Condition

SUMMARY:
BSA is a novel, computerized intervention specifically designed for active military personnel with the intent to reduce two risk factors known to be associated with suicide outcomes.

DETAILED DESCRIPTION:
The investigators have focused on the identification of malleable risk factors for preventative intervention in a number of types of psychopathology including suicidality. In the case of Perceived Burdensomeness (PB) and Thwarted Belongingness (TB), theory suggests that they may be malleable, though this has received little empirical attention. Taken together, the Interpersonal Theory of Suicide and related empirical literature suggest that targeting PB/TB should offer a novel and important avenue to reduce suicidality. This inspired the investigators' efforts to create and evaluate an intervention - called Building Stronger Allies (BSA) - designed to reduce these factors.

ELIGIBILITY:
Inclusion Criteria:

* Must show at least some suicide risk based on scoring > 0 on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Must also own a Smartphone.

Exclusion Criteria:

* No evidence of such serious suicidal risk that would indicate a need for immediate hospitalization or emergency intervention.
* No planned moves/deployments for the next 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Acquired Capability for Suicide Scale - Fearlessness About Death (ACSS-FAD) | Up to year three of the study
  7-item measure that assesses the degree to which individuals feel fearless or unafraid about death (Ribeiro et al., 2014).
Suicide Bereavement (ASF) | Up to year three of the study
  1 item created by the MSRC to obtain information regarding the experience of knowing someone who died by suicide.
Beck Suicide Scale (BSS) | Up to year three of the study
  21-item measure assessing a broad spectrum of behaviors and attitudes related to suicide risk, including suicidal ideation and past suicide attempts (Beck et al.,1979)
Depression Symptom Index - Suicidality Subscale (DSI-SS) | Up to year three of the study
  4-item measure to assess the frequency and intensity of suicidal ideation and impulses (Joiner et al., 2002).
Reasons for Living Inventory (RFL) | Up to year three of the study
  current study will use 18 items (3 from each of the 6 subscales) from the 48-item measure of how important, to each respective participant, are common reasons individuals give for not committing suicide (Linehan et al., 1983).
Suicidal Behaviors Questionnaire - Revised (SBQ-R) | Up to year three of the study
  4-item measure assessing four dimensions of suicide (lifetime ideation and attempts, 12 month frequency of ideation, threat of suicidal behavior, and likelihood of suicidal behavior; Osman et al., 2001).
Suicide Attempt History (SHF) | Up to year three of the study
  6 items created by the MSRC to assess history of suicide attempts, most lethal attempt, and non-suicidal self-injury.
Suicide Intensity Ratings (SIR) | Up to year three of the study
  3 items to assess current intent and desire to die by suicide, as well as current intensity of suicidal ideation.
Suicide Intent Questions (SIS) | Up to year three of the study
  4 items picked by the MSRC to assess thoughts and feelings during most recent engagement in self-injury with intent to die.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to year three of the study
  a structured clinical interview that measures the presence, frequency, and characteristics of various types of suicidal thoughts and behaviors.
Implicit Association Task (IAT) for Suicide | Up to year three of the study
  We will use Nock's IAT for suicide as a behavioral index of suicide risk. This procedure has demonstrated that implicit associations for death
  /self are stronger among those with a suicide attempt history relative to psychiatric controls without a history of suicide attempts.
Affect Misattribution Procedure (AMP) for Suicide | Up to year three of the study
  We will use a modified version of the AMP task using suicide-relevant stimuli as an additional implicit measure of suicide risk. A variant of this task has been found to predict suicidal behavior

SECONDARY OUTCOMES:
Attentional Control Scale (ACS) | Up to year three of the study
  20-item measure that assesses the differences in voluntary attentional control (Derryberry & Rothbart, 1988).
Anxiety Sensitivity Index - 3 (ASI-3) | Up to year three of the study
  18-item measure of anxiety sensitivity, or fears of anxiety related sensations (Taylor et al., 2007).
Anxiety and Stress Sensitivity (ASS) | Up to year three of the study
  26-item measure of anxiety, fear, or distress caused by a variety of symptoms or bodily sensations.
Alcohol Use Disorders Identification Test (AUDIT) | Up to year three of the study
  10-item measure of alcohol use and frequency of related problems or consequences (Saunders et al., 1993).
Beck Anxiety Inventory (BAI) | Up to year three of the study
  21-item measure of general anxiety symptomatology (Beck et al.,1988).
Beck Depression Inventory (BDI-II) | Up to year three of the study
  21-item measure that assesses severity of depressive symptomatology (Beck et al., 1988).
Beck Hopelessness Scale (BHS) | Up to year three of the study
  current study will use 3 of the 20 items in this measure to assess hopelessness (Beck et al., 1974)
Buss-Perry Aggression Questionnaire - Anger Subscale (BPAQ) | Up to year three of the study
  current study will use the 7-item anger subscale of this 29-item measure to assess participant's experience and expression of anger (Buss & Perry, 1992)
Centers for Disease Control and Prevention Behavioral Risk Factor Surveillance System State (BRFSS) | Up to year three of the study
  3-item measure about possession of firearms.
Client Expectancy Questionnaire (CEQ) | Up to year three of the study
  8-item questionnaire measuring treatment expectancy and rationale credibility for use in clinical outcome studies (Devilly & Borkovec, 2000).
Client Satisfaction Questionnaire (CSQ) | Up to year three of the study
  8-item measure assessing general satisfaction with services of treatment received by the individual (Attkisson & Zwick, 1982)
DARTS Quiz | Up to year three of the study
  11-item measure assessing general satisfaction with an intervention by asking questions regarding presentation, applicability, and acceptability
Disturbing Dream and Nightmare Severity Index (DDNSI) | Up to year three of the study
  up to 16-item measure of nightmare severity and frequency (Krakow et al., 2002)
Demographics | Up to year three of the study
  scale was created to collect data on the participants' gender, ethnicity, educational/occupational level, and current medications. It includes additional questions about military service career variables (e.g., duration of active duty, number of deployments).
Drug Use Questions (DUQ) | Up to year three of the study
  2 items created by the MSRC to assess frequency of prescription medication abuse and non-prescription/recreational drug use
Dyadic Adjustment Scale (DAS) | Up to year three of the study
  32-item measure of satisfaction in an intimate relationship (Spanier, 1976).
Engagement in Behavioral Health Treatment (EBHT) | Up to year three of the study
  1 item created by the MSRC to assess number of behavioral health treatment sessions attended in the previous 3 months.
Interpersonal Needs Questionnaire (INQ-R) | Up to year three of the study
  15-item measure of the constructs of thwarted belongingness and perceived burdensomeness as defined by the Interpersonal Theory of Suicide (Van Orden et al., 2012).
*Insomnia Severity Index (ISI) | Up to year three of the study
  7-item measure of the symptoms of and consequences of insomnia and the degree of concerns/distress caused by those difficulties (Bastien et al., 2001).
Positive and Negative Affect Scale - Negative Affect Subscale (PANAS-NA) | Up to year three of the study
  10-item measure of levels of negative affect (Watson et al., 1988).
PTSD Checklist for DSM-5 (PCL-5) | Up to year three of the study
  20-item measure of symptoms of PTSD (Blevins et al., 2015).
Relationship Closeness Inventory (RCI) | Up to year three of the study
  measure of interpersonal closeness in a relationship (Snyder & Omoto, 1989). It consists of three subscales assessing amount of time spent together (Frequency), number of different activities done together (Diversity), and the influence another has on one's behaviors, activities, and decisions (Strength)
Sheehan Disability Scale (SDS) | Up to year three of the study
  4-item measure assessing degree of impairment and disability in several main life areas (Sheehan, 1983)
Social Interaction Anxiety Scale (SIAS) | Up to year three of the study
  20-item measure assessing fears of general social interactions (Mattick & Clarke, 1998).
Traumatic Brain Injury - 4 (TBI-4) | Up to year three of the study
  4-items to screen for potential traumatic brain injuries (Brenner et al., 2012).
Use of Behavioral Health Services (UBHS) | Up to year three of the study
  2 items created by the MSRC to assess the effects of psychotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lora R Hunter, PhD, Study Chair — Medical Service Corps, United States Army
Locations (1):
- 101st Airborne Division (Air Assault) Combat Aviation Brigade, Fort Campbell North, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No